CLINICAL TRIAL: NCT02883647
Title: Clinical Investigation About Therapeutic Effects and Long-term Follow-up After Ending Anti-hepatitis B Virus Therapy With Nucleos(t)Ide Analogs in Patients With Chronic Hepatitis b
Brief Title: Therapeutic Effects and Long-term Follow-up After Ending Nucleos(t)Ide Analogs Therapy in Chronic Hepatitis b
Status: Recruiting | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Associated Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: PL
Record Dates: First submitted 2016-06-13; First posted 2016-08-30 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hepatitis b
Keywords: chronic hepatitis b, nucleos(t)ide analog
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- retreatment: 1. Patients with HBV DNA > 2000 IU/ml and ALT ≥ 5×ULN;
  2. Patients with HBV DNA > 2000 IU/ml and 2×ULN < ALT ≤ 5×ULN, but have clinical symptoms.
  Intervention: Patients of this group will receive Entecavir 0.5mg/d or Tenofovir 300mg/d again.
  Interventions: Drug: Entecavir or Tenofovir
- non-retreatment: 1. Patients with HBV DNA ≤ 2000 IU/ml;
  2. Patients with HBV DNA > 2000 IU/ml and ALT ≤ 2×ULN;
  3. Patients with HBV DNA > 2000 IU/ml and 2×ULN < ALT ≤ 5×ULN, but have no clinical symptoms.

INTERVENTIONS:
Drug: Entecavir or Tenofovir — Patients in retreatment group receive nucleos(t)ide analogs therapy (Entecavir 0.5mg/d or Tenofovir 300mg/d) again
  Groups: retreatment

SUMMARY:
The study is to observe the therapeutic effects and long-term follow-up after ending anti-HBV therapy with nucleos(t)ide analogs in patients with chronic hepatitis b.

DETAILED DESCRIPTION:
Patients with chronic hepatitis b were enrolled in the study. Age, sex, weight, height, symptoms (e.g., fatigue, poor appetite, jaundice), relapse, retreatment, occurrence of liver cirrhosis and hepatocellular carcinoma (HCC), mortality and survival rate were recorded in the study. We also observed the laboratory tests including the levels of white blood cells (WBC), red blood cells (RBC), hemoglobin (HGB), platelet (PLT), alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin (TBIL), blood urea nitrogen (BUN), creatine, hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), hepatitis B virus (HBV) DNA, CD4 positive T lymphocyte (CD4+T), CD8 positive T lymphocyte (CD8+T), Type 1 helper T lymphocyte (Th1), Type 2 helper T lymphocyte (Th2),fibroscan and B ultrasound. If clinical relapse occurred, patients were retreated with nucleos(t)ide analogs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients received anti-HBV therapy with nucleos(t)ide analogs.
2. Last anti-HBV therapy should continue for at least 2 years.
3. For HBeAg positive patients, HBV DNA should keep negative for at least 1 year after HBeAg seroconversion before the therapy ending; for HBeAg negative patients, HBV DNA should keep negative for at least 2 years before the therapy ending.

Exclusion Criteria:

1. Liver cirrhosis, HCC;
2. Patients with other factors causing active liver diseases;
3. Pregnancy or lactation;
4. Patients with HIV infection or congenital immune deficiency diseases;
5. Patients with severe diabetes, autoimmune diseases, other important organ dysfunctions and other serious complications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of chronic hepatitis b
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01-01; Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
relapse | up to 48 weeks
  non-relapse:serum HBV DNA < 2000 IU/ml; virologic relapse: serum HBV DNA > 2000 IU/ml; clinical relapse:serum HBV DNA > 2000 IU/ml and ALT > 2×ULN

SECONDARY OUTCOMES:
occurence of cirrhosis and hepatocellular carcinoma | up to 48 weeks
  sign of cirrhosis and hepatocellular carcinoma through ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wu L, Lai J, Luo Q, Zhang Y, Lin C, Xie D, Chen Y, Deng H, Gao Z, Peng L, Xu W. Long-term hepatitis B surface antigen kinetics after nucleos(t)ide analog discontinuation in patients with noncirrhotic chronic hepatitis B. Liver Res. 2024 Jul 6;8(3):179-187. doi: 10.1016/j.livres.2024.07.001. eCollection 2024 Sep. PMID 39957751
- [Derived] Xu WX, Zhang Q, Zhu X, Lin CS, Chen YM, Deng H, Mei YY, Zhao ZX, Xie DY, Gao ZL, Xie C, Peng L. 48-Week Outcome after Cessation of Nucleos(t)ide Analogue Treatment in Chronic Hepatitis B Patient and the Associated Factors with Relapse. Can J Gastroenterol Hepatol. 2018 May 10;2018:1817680. doi: 10.1155/2018/1817680. eCollection 2018. PMID 29862225